CLINICAL TRIAL: NCT03633552
Title: A Single-blind, Randomized, Clinical Trial Comparing the Efficacy of 6 Cycles Versus 12 Cycles Temozolomide Regimens in Adjuvant Treatment of Patients With Brain High Grade Glioma
Brief Title: Efficacy of Two Temozolomide Regimens in Adjuvant Treatment of Patients With Brain High Grade Glioma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyed Alireza Javadinia, Principal Investigator, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 960021; IRCT20160706028815N3 (Registry Identifier: Iranian Registry of Clinical Trials)
Record Dates: First submitted 2018-07-20; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Glioblastoma Multiforme of Brain; Anaplastic Astrocytoma of Brain
Keywords: Glioblastoma Multiforme; Anaplastic Astrocytoma; Adjuvant treatment; Extended chemotherapy
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: The patients will be randomized to 6-cycle and 12-cycle adjuvant Temozolomide groups using block randomization method (1:1).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 12-cycle arm (Experimental): After completion of chemoradiation, the cases will receive 12 cycles of adjuvant Temozolomide (prescribed as 150 to 200 milligram per square meters body surface per day for the first 5 days of every 28 days).
  Interventions: Drug: Temozolomide
- 6-cycle arm (Active Comparator): After completion of chemoradiation, the participants will receive 6 cycles of adjuvant Temozolomide (prescribed as 150 to 200 milligram per square meters body surface per day for the first 5 days of every 28 days).
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — The patients will initially undergo surgery. Within 4 to 6 weeks after surgery, all patients will receive chemoradiation. After completion of chemoradiation, the cases will receive 12 cycles of adjuvant Temozolomide (prescribed as 150 to 200 milligram per square meter body surface per day for the first 5 days of every 28 days). In the control group, the patients will receive 6 cycles of adjuvant Temozolomide (in the same dosage).
  Other Names: Temodar, Temodal, Temcad, Glidar

SUMMARY:
This is a phase III, non-blinded, blocked randomized clinical trial. The study is conducted on 62 newly diagnosed patients with brain glioblastoma multiforme and anaplastic astrocytoma referring to the oncology clinics during March 2018 and March 2019. The patients will be randomized to 6-cycle and 12-cycle adjuvant Temozolomide groups using block randomization method (1:1).

DETAILED DESCRIPTION:
This study aimed to compare the overall survival and progression free survival between 6 cycles and 12 cycles adjuvant Temozolomide regimens in patients with brain glioblastoma and anaplastic astrocytoma. The main inclusion criterion includes patients newly diagnosed with glioblastoma and anaplastic astrocytoma whose diagnosis is confirmed by histologic evaluation. The main exclusion criteria involve chronic renal, hepatic or cardiac failure. The patients will initially undergo surgery. Within 4 to 6 weeks after surgery, all patients will receive chemoradiation. After completion of chemoradiation, the cases will receive 12 cycles of adjuvant Temozolomide (prescribed as 150 to 200 milligram per square meter body surface per day for the first 5 days of every 28 days). In the control group, the patients will receive 6 cycles of adjuvant Temozolomide (in the same dosage). This is a phase III, non-blinded, blocked randomized clinical trial. The study is conducted on 62 newly diagnosed patients with brain glioblastoma multiforme and anaplastic astrocytoma referring to the oncology clinics during March 2018 and March 2019. The patients will be randomized to 6-cycle and 12-cycle adjuvant Temozolomide groups using block randomization method (1:1). This study will be conducted in the oncology clinic of Omid Hospital and Imam Reza Hospital, Mashhad. Blinding is not observed in this study. The primary endpoints of study are overall survival and progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed glioblastoma and anaplastic astrocytoma
* age between 18 and 70 years
* Karnofsky Performance Scale Index equal or more than 60 percent
* signed informed consent

Exclusion Criteria:

* chronic hepatic
* renal failure
* cardiac failure
* history of hematologic malignancies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-03-03 (Actual); Primary Completion 2021-03-03 (Estimated); Study Completion 2021-04-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 1 year from start of treatment
  The time interval between the diagnosis and death.
Progression-free survival | up to 1 year from start of treatment
  The time interval between the diagnosis and disease progression based on radiologic criteria or symptoms

SECONDARY OUTCOMES:
Anemia | monthly, up to 12 months during treatment
  blood hemoglobin lower than 10 grams per deciliter
Neutropenia | monthly, up to 12 months during treatment
  Blood almost mature neutrophils count lower than 1500/mm3
Presence of alopecia | monthly, up to 12 months during treatment
  A condition in which hair is lost
Presence of nausea | monthly, up to 12 months during treatment
  An unpleasant sense of unease, discomfort, and revulsion towards food
Presence of vomiting | monthly, up to 12 months during treatment
  Eject matter from the stomach through the mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Mahdi Silanian Toosi, M.D., Study Director — Mashhad University of Medical Sciences; Kazem Anvari, M.D., Study Chair — Mashhad University of Medical Sciences
Locations (2):
- Iran (2):
  - Radiation ward of Emam Reza Hospital, Mashhad, Razavi Khorasan Province
  - Omid Hospital, Mashhad, Razavi Khorasan Province

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make this available.